CLINICAL TRIAL: NCT02348957
Title: Treating Patients With Chronic Myeloid Leukemia (CML) in Chronic Phase (CP) With Dasatinib PCR-Monitoring, Adherence, Quality of Life, Therapy Satisfaction
Brief Title: Treating Patients With Chronic Myeloid Leukemia (CML) in Chronic Phase (CP) With Dasatinib
Acronym: DasPAQT
Status: Completed | Type: Observational
Sponsor: Onco Medical Consult GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: OMC 2014-I
Record Dates: First submitted 2014-12-15; First posted 2015-01-28 (Estimated); Last update posted 2019-07-25 (Actual); Status verified 2018-07

CONDITIONS: Myeloid Leukemia, Chronic, Chronic-Phase
Keywords: Chronic myeloid leukemia; Dasatinib; Any line; Chronic phase
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
CML requires ongoing treatment and assessment of treatment milestones in order to manage the disease properly. Dasatinib is approved for the treatment of newly diagnosed PH+ CP-CML and CML in chronic or accelerated phase or blast crisis in patients resistant or intolerant to prior therapies including Imatinib. Although Imatinib has demonstrated unprecedented efficacy in clinical trials, mostly in chronic phase CML, there is lack of published data on how CML is managed in real-life clinical practice settings. Therefore this non-interventional study is designed to collect real-life data on CML-treatment with Dasatinib in clinical routine with respect to first and second line treatment and/or switch setting (within 1st line or from 1st line TKI to 2nd line Dasatinib). Emphasis lies on health care provided in registered doctor's practices as here most of CML patients who are not involved in clinical trials are treated.

DETAILED DESCRIPTION:
The advent of Imatinib into the market in 2001 changed the treatment paradigm of CML. Seven-year follow-up from the IRIS trial revealed an estimated overall survival of 86% in newly diagnosed CML patients treated with Imatinib.

In June 2006, the U.S. Food and Drug Administration (FDA) granted accelerated approval for Dasatinib to treat adults with CP-CML with resistant disease or who were intolerant to prior therapy, including Imatinib. The FDA converted Dasatinib to a regular approval in May 2009, after confirmation of the treatment's safety and effectiveness. On October 28, 2010, FDA granted accelerated approval to Dasatinib for the treatment of newly diagnosed adult patients with CML-CP. Dasatinib entered thereby a marketplace with other TKIs including Nilotinib.

According to the summary of product characteristics brochure Dasatinib (Sprycel®) is indicated for the treatment of adult patients with:

* Newly diagnosed Ph+ CML In the chronic phase.
* Chronic, accelerated or blast phase CML with resistance or intolerance to prior therapy including Imatinib mesilate.
* Ph+ acute lymphoblastic leukaemia and lymoid blast CML with resistance or intolerance to prior therapy.

A phase III study (DASISION) of Dasatinib vs. Imatinib could proof that Dasatinib induced significantly higher and faster rates of complete cytogenetic response and major molecular response when compared to Imatinib. Since achieving complete cytogenetic response within 12 months has been associated with better long-term, progression-free survival, Dasatinib may improve the long-term outcomes among patients with newly diagnosed chronic-phase CML.

Nevertheless, further data are required to obtain additional information on the clinical benefits of Dasatinib.

CML requires ongoing treatment and assessment of treatment milestones in order to manage the disease properly. Dasatinib is approved for the treatment of newly diagnosed PH+ CP-CML and CML in chronic or accelerated phase or blast crisis in patients resistant or intolerant to prior therapies including Imatinib. Although Imatinib has demonstrated exceptional efficacy in clinical trials, mostly in chronic phase CML, there is lack of published data on how CML is managed in real-life clinical practice settings.

Therefore this non-interventional study is designed to collect real-life data on CML-treatment with Dasatinib in clinical routine with respect to first and second line treatment and/or switch setting (within 1st line or from 1st line TKI to 2nd line Dasatinib). Emphasis lies on health care provided in registered doctor's practices as here most of CML patients who are not involved in clinical trials are treated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed CP-CML and CML patients in chronic phase resistant or intolerant to prior therapies, including Imatinib. Any line treatment of chronic CML.
* 18 years or older at time of diagnosis
* Receiving treatment with Dasatinib according to the SmPC
* Written informed consent obtained before any screening procedure and according to local guidelines

Exclusion Criteria:

•Patients who are participating in a clinical trial for CML treatment will be excluded

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This non-interventional study will document around 300 adult patients with newly-diagnosed CP-CML and CML patients in chronic phase resistant or intolerant to prior therapies, including Imatinib and Nilotinib.
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2014-10; Primary Completion 2019-03 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Distribution of Molecular remission status at study entry and after 12 months. | 12 Months
  Patients included into this study are on a treatment with Dasatinib. Fraction of BCR-ABL positive cells is measured at study entry or was assessed at the timepoint of Dasatinib treatment begin and classified as >MR3, MR3, MR4, and MR4.5 as an ordinal measure.
  Molecular Fraction of BCR-ABL positive cells is reassessed after 12 months.

SECONDARY OUTCOMES:
Distribution of Molecular remission status at study entry and after 24 months. | 24 months
  Patients included into this study are on a treatment with Dasatinib. Fraction of BCR-ABL positive cells is measured at study entry or was assessed at the time point of Dasatinib treatment begin and classified as >MR3, MR3, MR4, and MR4.5 as an ordinal measure.
  Molecular Fraction of BCR-ABL positive cells is reassessed after 24 months.
Best possible response | Up to 36 months
  Defined as the best response at any time after the start of the treatment. Reported will be distributions for each response (progression, stable disease, remission for at least one class of MR)
Time to Molecular remission | up to 36 months
  Patients reach this event, when a change from a higher amount of BCR-ABL positive patients to a lower amount of BCR-ABL positive patients occurs
Time molecular progression | Up to 36 months
  Patients start the observation period at study entry and reach this event, when a change to a higher BCR-ABL remission status is reached.
Cytogenetic profile at start of Dasatinib treatment, type of BCR-ABL transcript (if these parameters are routinely tested at the facility and are documented for the NIS). | Up to 36 months
  Cytogenetic response according to conventional cytogenetics (evaluation of at least 20 metaphase chromosomes) and hyper metaphase FISH (if applicable)
Hematologic response (HR) and complete blood count (if these parameters are routinely tested at the facility and are documented for the NIS) | Up to 36 months
  Complete blood count (if these parameters are routinely tested at the facility and are documented for the NIS
Patient Compliance/Adherence | After 3,6,12,24 months
  Assessed at Baseline and analyzed over time after 3,6,12,24 months of observation.
Patients' Satisfaction | After 3,6,12,24 months
  Assessed at Baseline and analyzed over time after 3,6,12,24 months of observation.
Quality of Life | Time after 3,6,12,24 months
  Assessed at Baseline and analyzed over time after 3,6,12,24 months of observation.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Time after 3,6,12,24 months
  Assessed at Baseline and analyzed over time after 3,6,12,24 months of observation.
Subgroup analysis concerning the primary study objective | 12 months
  Common influencing factors like prognostic scores or previous therapy patterns are analyzed, whether they have an influence on the primary study aim.
Subgroup analysis concerning the time to remission | Up to 36 months
  Common influencing factors like prognostic scores or previous therapy patterns are analyzed, whether they have an influence on time to remission
Subgroup analysis concerning the time to progression | Up to 36 months
  Common influencing factors like age, sex or previous therapy patterns are analyzed, whether they have an influence on time to progression
Subgroup analysis concerning the quality of life and patient compliance | Time after 3,6,12,24 months
  Common influencing factors like age, sex, comorbidities or previous therapy patterns are analyzed, whether they have an influence on quality of life and patient compliance
Subgroup analyses of participants with Adverse Events as a Measure of Safety and Tolerability | Time after 3,6,12,24 months
  Common influencing factors like age, sex, comorbidities or previous therapy patterns are analyzed, whether they have an influence on safety and toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Hans Tesch, Prof. Dr., Principal Investigator — Hämatologisch-Onkologische Gemeinschaftspraxis am Bethanien-Krankenhaus, Im Prüfling 17, D-60389 Frankfurt am Main
Locations (66):
- Germany (66):
  - Praxis für Hämatologie und internistische Onkologie, Heidenheim, Baden-Wurttemberg
  - Ambulantes Therapiezentrum, Offenburg, Baden-Wurttemberg
  - Diakonie-Klinikum Schwäbisch Hall GmbH, Klinik für Innere Medizin III, Schwäbisch Hall, Baden-Wurttemberg
  - Praxisklinik für integrative Onkologie, Altötting, Bavaria
  - Gemeinschaftspraxis Drs. Klausmann, Aschaffenburg, Bavaria
  - Klinikum Aschaffenburg Hämato-Onkologische Schwerpunktpraxis, Aschaffenburg, Bavaria
  - Onkologische Gemeinschaftspraxis, Bamberg, Bavaria
  - Klinikum Bayreuth Klinik für Hämatologie und Onkologie, Bayreuth, Bavaria
  - Schwerpunktpraxis für Hämatologie und Onkologie, Bayreuth, Bavaria
  - Onkologische Schwerpunktpraxis, Kronach, Bavaria
  - Hämatologie Onkologie Palliativmedizin Tagesklinik Landshut, Landshut, Bavaria
  - Facharztpraxis für Hämatologie und Onkologie, München, München, Bavaria
  - Praxis für Hämatologie und Onkologie am Isartor, München, Bavaria
  - MOP-Studiengesellschaft, München, Bavaria
  - Schwerpunktpraxis und Tagesklinik dür Hämatologie und Onkologie/OncoPRO GbR, Regensburg, Bavaria
  - Fachärztliche Gemeinschaftspraxis, Weiden, Bavaria
  - MVZ für Blut- und Krebserkrankungen Potsdam, Potsdam, Brandenburg
  - Onkologische Schwerpunktpraxis und Tagesklinik, Bad Soden am Taunus, Hesse
  - Onkologische Gemeinschaftspraxis am Bethanien-Krankenhaus, Frankfurt am Main, Hesse
  - Gemeinschaftspraxis Dres med. Dirk Meyer & Andreas Ammon und Michael Metz, Göttingen, Hesse
  - Onkologische Schwerpunktpraxis, Hanau, Hesse
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Langen, Hesse
  - Dres. Klaus Maria Josten und Ortwin Klein, Wiesbaden, Hesse
  - Onkologische Kooperation Harz, Goslar, Lower Saxony
  - Onkologisches Ambulanzzentrum Hannover, Hanover, Lower Saxony
  - Praxis für Hämatologie und Onkologie, Hanover, Lower Saxony
  - Onkologische Schwerpunktpraxis Hildesheim, Hildesheim, Lower Saxony
  - Schwerpunktpraxis, Neustadt am Rübenberge, Lower Saxony
  - Intern. Gemeinschaftspraxis, Güstrow, Mecklenburg-Vorpommern
  - Gemeinschaftspraxis für Hämatologie/Onkologie, Rostock, Mecklenburg-Vorpommern
  - Hämatologisch-onkologische Gemeinschaftspraxis Nordhorn, Nordhorn, Niedersachen
  - MVZ Arnsberg, Arnsberg, North Rhine-Westphalia
  - Vinzenz Pallotti Hospital GmbH, Bergisch Gladbach, North Rhine-Westphalia
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Cologne, North Rhine-Westphalia
  - Gemeinschaftspraxis für Hämatologie und Onkologie / Ambulante Tumortherapie, Cologne, North Rhine-Westphalia
  - Medizinisches Versorgungszentrum (MVZ) an der St. Marien-Hospital Düren gGmbH, Düren, North Rhine-Westphalia
  - Onko.Logix GmbH & Co. KG, Gelsenkirchen, North Rhine-Westphalia
  - Praxis für Hämatologie und Onkologie, Hamm, North Rhine-Westphalia
  - Praxisklinik Hämatologie/Onkologie Herne, Herne, North Rhine-Westphalia
  - Klinikum Lippe Onkologie und Hämatologie, Lemgo, North Rhine-Westphalia
  - Praxis für Hämatologie, Onkologie und Palliativmed, Mönchengladbach, North Rhine-Westphalia
  - Onkologische Schwerpunktpraxis Mülheim an der Ruhr und Oberhausen, Mülheim, North Rhine-Westphalia
  - Onkologische Praxis Remscheid, Remscheid, North Rhine-Westphalia
  - Klinikum Idar-Oberstein GmbH Medizinische Klinik I, Idar-Oberstein, Rhineland-Palatinate
  - IDGGQ, Institut für med. Dokumentation GbR, Kaiserslautern, Rhineland-Palatinate
  - Praxisklinik für Hämatologie und Onkologie Koblenz/ Institut für Versorgungsforschung in der Onkologie GbR, Koblenz, Rhineland-Palatinate
  - CaritasKlinikum Saarbrücken St. Theresia Akademisches Lehrkrankenhaus der Universität des Saarlandes, Saarbrücken, Saarland
  - Gemeinschaftspraxis Drs. Georg Jacobs, Prof Heiner Daus und PD Dr. Schmits, Saarbrücken, Saarland
  - Onkologische Praxis Bautzen, Bautzen, Saxony
  - Klinikum Chemnitz gGmbH Klinik für Innere Medizin III, Chemnitz, Saxony
  - Internistische Praxis & Tagesklinik, Neustadt, Saxony
  - Ambulante Onkologie Ostsachsen, Zittau, Saxony
  - Hämato-onkologische Praxis, Halberstadt, Saxony-Anhalt
  - Gemeinschaftspraxis, Eisenach, Thuringia
  - Onkologische Schwerpunktpraxis Augsburg, Augsburg
  - OVZ Friedrichshain Hämatologie, Onkologie und Palliativmedizin, Berlin
  - Krebsheilkunde Lichtenberg, Berlin
  - Praxis für Innere Medizin Ärztehaus Berlin-Pankow, Berlin
  - Medizinische Klinik mit Schwerpunkt Hämatologie, Onkologie und Tumorimmunologie Charité - Universitätsmedizin Berlin, Berlin
  - Onkologie Duisburg Nord, Duisburg
  - Onkologie Lerchenfeld, Hamburg
  - Onkologie Hof - Medizinisches Versorgungszentrum GmbH, Hof
  - Hämatologische Praxisgemeinschaft München, München
  - Schwerpunktpraxis für Hämatologie und Internistische Onkologie, Gastroenterologie, Singen
  - Onkologische Schwerpunktpraxis Trier St. Anna / Brüderkrankenhaus, Trier
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Westerstede